CLINICAL TRIAL: NCT07097701
Title: An Open-Label, Randomized, Cross-Over Study to Investigate the Efficacy and Safety of Mexiletine PR Compared to Mexiletine IR in Patients With Non-Dystrophic Myotonias (ACHILLES Study)
Brief Title: An Open-Label, Randomized, Cross-Over Study to Investigate the Efficacy and Safety of Mexiletine PR Compared to Mexiletine IR
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Lupin Ltd. (Industry)
Collaborators: Lupin Atlantis Holdings S.A. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: MEX-NDM-301
Record Dates: First submitted 2024-11-21; First posted 2025-07-31 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Myotonia
MeSH Terms: conditions — Myotonia | interventions — Mexiletine

STUDY DESIGN:
Intervention Model Description: This is a multicenter, open-label, randomized, cross-over study intended to evaluate the efficacy and the safety of mexiletine PR (QD) vs mexiletine IR (TID) in patients with non-dystrophic myotonias including myotonia congenita (MC), paramyotonia congenita (PC) and sodium channel myotonia (SCM). The study will consist of a 4-week screening period followed by two 12-week treatment periods. Eligible patients will be randomized to receive mexiletine PR or mexiletine IR for 12 weeks. After a wash out period of at least 7 days the patients will receive the opposite treatment for 12 weeks.
  A total of 24 patients are planned to be enrolled (with a target enrollment of 12 naïve to previous mexiletine treatment and 12 previously treated with mexiletine).
Who Masked: Participant
Masking Description: Study drug (mexiletine PR or mexiletine IR) will be started as a 167 mg once a day (QD) treatment regimen. The dose will be titrated up at Week 1 to 333 mg and at Week 2 to a maximum dose of 500 mg. All dose escalations will be done with safety ECG assessments using portable ECG device. Study drug should be taken at the beginning of the meal at approximately the same time of the day every day, preferably in the morning for Mexiletine PR or Mexiletine IR QD. Mexiletine IR twice a day (BID) should be taken in the morning and afternoon and Mexiletine IR TID should be taken in the morning, afternoon, and evening.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mexiletine prolonged-release (PR) (Active Comparator): Mexiletine PR 167 mg (mexiletine HCl 200 mg) Mexiletine PR 333 mg (mexiletine HCl 400 mg) OR Mexiletine PR 500 mg (mexiletine HCl 600 mg)
  Interventions: Drug: Granular powder in unit dose foil-lined sachet Mexiletine (PR)
- Mexiletine immediate release (IR) (Active Comparator): Mexiletine IR 167 mg (mexiletine HCl 200 mg)
  Interventions: Drug: Oral Capsule Mexiletine (IR)

INTERVENTIONS:
Drug: Granular powder in unit dose foil-lined sachet Mexiletine (PR) — Mexiletine (PR)
  Arms: Mexiletine prolonged-release (PR)
Drug: Oral Capsule Mexiletine (IR) — Mexiletine (IR)
  Arms: Mexiletine immediate release (IR)

SUMMARY:
An Open-Label, Randomized, Cross-Over Study to Investigate the Efficacy and Safety of Mexiletine PR compared to Mexiletine IR in Patients with Non-Dystrophic Myotonias (ACHILLES study)

DETAILED DESCRIPTION:
This is a multicenter, open-label, randomized, cross-over study intended to evaluate the efficacy and the safety of mexiletine PR (QD) vs mexiletine IR (TID) in patients with non-dystrophic myotonias including myotonia congenita (MC), paramyotonia congenita (PC) and sodium channel myotonia (SCM). The study will consist of a 4-week screening period followed by two 12-week treatment periods. Eligible patients will be randomized to receive mexiletine PR or mexiletine IR for 12 weeks. After a wash out period of at least 7 days the patients will receive the opposite treatment for 12 weeks.

A total of 24 patients are planned to be enrolled (with a target enrollment of 12 naïve to previous mexiletine treatment and 12 previously treated with mexiletine).

Safety assessments include patient- and physician-reported adverse event reporting, electrocardiogram (ECG), standard clinical laboratory evaluations, physical examinations, and vital signs. Efficacy assessments include patient-reported outcomes (PROs) and functional capacity outcome measures.

ELIGIBILITY:
Inclusion Criteria

1. Ability to comprehend and willingness to sign an informed consent (ICF) or ICF of the parent(s)/legal guardian and written assent from the patient (if patient < 18 years of age);
2. Non-dystrophic myotonias including myotonia congenita (MC), paramyotonia congenita (PC) and sodium channel myotonia (SCM) confirmed genetically;
3. Male or non-pregnant female ≥16 years and older at screening;
4. Body Mass Index (BMI) of 18.5 kg/m2 to 30 kg/m2, and weight ≥45 kg;
5. Female patients of childbearing potential must be using a highly effective form of birth control for the duration of the study and for at least 30 days after last dose of study drug. Male patients must use birth control for the duration of the study and for at least 30 days after last dose of study drug;
6. No significant cardiac abnormalities as determined by a cardiologist including electrocardiogram (ECG) and echocardiogram not older than 3 months prior to study entry;
7. Participants with myotonic symptoms severe enough to justify treatment (in the opinion of the study investigator);
8. Presence of clinical handgrip myotonia (delayed relaxation of grip of ≥ 3 second using a stopwatch) at screening (naïve patients only) and on Day 1 (pre-dose) (patients naïve and previously treated with mexiletine).

Exclusion Criteria

1. Are pregnant or lactating;
2. Have any one of the following medical conditions: uncontrolled diabetes mellitus, cancer other than skin cancer less than five years previously (e.g., basal-cell carcinoma (BCC) and squamous-cell carcinoma (SCC) of skin allowed), multiple sclerosis, seizure disorders, or other serious medical illness or has any other condition, which in the opinion of the Investigator, precludes the participant's participation in the study or the participant is unlikely to comply with the protocol-defined procedures and therefore is unlikely to complete the study;
3. Severe renal impairment (glomerular filtration rate (GFR) < 30 mL/min);
4. Medical conditions which could interfere with muscle function such as infections, trauma, fractures, or planned surgery;
5. Medical conditions that could affect hand functioning including but not limited to rheumatoid arthritis, Dupuytren's contracture, hand deformity, etc.;
6. Severe arthritis or medical condition (other than NDM) that would significantly impact ambulation;
7. Severe hepatic impairment or preexisting elevated liver function tests > 3 times the upper limit of normal (ULN) at screening (alanine transaminase (ALT)/aspartate transaminase (AST), gamma-glutamyl transferase (GGT)) and/or any abnormal chemistry, hematology or urine lab considered clinically significant by the investigator;
8. Serum potassium values < 3.5 mmol/L or > 5.0 mmol/L or serum magnesium values < 1.7 mg/dL. Electrolytic imbalance such as hypocalcaemia, hypercalcaemia, hypokalaemia, hyperkalaemia or hypomagnesaemia may increase the proarrhythmic effects of mexiletine. Electrolyte imbalances need to be corrected before administering mexiletine and will be monitored throughout treatment.
9. Intake of any other anti-myotonic treatment within 4 weeks prior to baseline (Day 1) or 5 half-lives, whichever is longer (e.g., metformin, propafenone, flecainide, lamotrigine, carbamazepine or any other channel-blocker/anticonvulsive drugs;
10. Use of any concomitant medications that could increase the cardiac risk or increases the risk of adverse reactions (see Section 6.8 for a complete list of prohibited concomitant medications);
11. Known allergy to mexiletine or any of the excipients or any local anesthetics;
12. Participation in another interventional clinical study during the last 3 months or 5 half-lives of the investigational medicinal product, whichever is longer;
13. Wheelchair-bound or bedridden;
14. Any cardiac safety-associated condition including any of the following criteria detected by screening cardiac evaluations including ECG, echocardiogram and clinical evaluations (see protocol Section 5.3 for a detailed list);
15. Current smokers (within one month of the screening visit) (eg, cigarettes, cigars, vape/e-cigarette products, etc.);
16. Subgroup 'mexiletine-naïve': patients with previous treatment with mexiletine are excluded. Subgroup 'previous mexiletine treatment': patients with treatment with mexiletine within 1 week prior to baseline (Day 1) are excluded

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-09-03 (Actual); Primary Completion 2027-01-22 (Estimated); Study Completion 2027-02-22 (Estimated)

PRIMARY OUTCOMES:
To compare the safety of mexiletine PR vs mexiletine IR by incidence of treatment emergent Adverse Events (TEAEs), treatment-related TEAEs, serious AEs, and patient discontinuation rate between mexiletine PR and mexiletine IR after 12 weeks of treatment. | Baseline to week 24
  To compare the safety of mexiletine PR vs mexiletine IR for the symptomatic treatment of myotonia in adult patients with non-dystrophic myotonias (myotonia congenita (MC), paramyotonia congenita (PC) and sodium channel myotonia (SCM)) by incidence of treatment emergent Adverse Events (TEAEs), treatment-related TEAEs, serious AEs, and patient discontinuation rate between mexiletine PR and mexiletine IR after 12 weeks of treatment.
To compare the safety of mexiletine PR vs mexiletine IR by mean change from baseline in QTc intervals by12-lead in ECG | Baseline to week 24
  To compare the safety of mexiletine PR vs mexiletine IR for the symptomatic treatment of myotonia in adult patients with non-dystrophic myotonias (myotonia congenita (MC), paramyotonia congenita (PC) and sodium channel myotonia (SCM)) by mean change from baseline in QTc Intervals by12-lead in ECG
To compare the safety of mexiletine PR vs mexiletine IR by mean change from baseline in PR intervals by12-lead in ECG | Baseline to week 24
  To compare the safety of mexiletine PR vs mexiletine IR for the symptomatic treatment of myotonia in adult patients with non-dystrophic myotonias (myotonia congenita (MC), paramyotonia congenita (PC) and sodium channel myotonia (SCM)) by mean change from baseline in PR intervals by12-lead in ECG.
To compare the safety of mexiletine PR vs mexiletine IR by mean change from baseline in QRS intervals by12-lead in ECG | Baseline to week 24
  To compare the safety of mexiletine PR vs mexiletine IR for the symptomatic treatment of myotonia in adult patients with non-dystrophic myotonias (myotonia congenita (MC), paramyotonia congenita (PC) and sodium channel myotonia (SCM)) by mean change from baseline in QRS intervals by12-lead in ECG
To compare the safety of mexiletine PR vs mexiletine IR by mean change from baseline by average minimum heart rate by12-lead in ECG | Baseline to week 24
  To compare the safety of mexiletine PR vs mexiletine IR for the symptomatic treatment of myotonia in adult patients with non-dystrophic myotonias (myotonia congenita (MC), paramyotonia congenita (PC) and sodium channel myotonia (SCM)) by mean change from baseline in average heart rate by 12-lead in ECG
To compare the safety of mexiletine PR vs mexiletine IR by performing physical examiniations | Baseline to week 24
  To compare the safety of mexiletine PR vs mexiletine IR for the symptomatic treatment of myotonia in adult patients with non-dystrophic myotonias (myotonia congenita (MC), paramyotonia congenita (PC) and sodium channel myotonia (SCM)) by performing physical examinations. The investigator will complete a physical examination including the following regions and systems: general appearance, head and neck, heart, lung, abdomen, chest and back, upper extremities, lower extremities, neurological, and dermatological. In addition, height and weight will be recorded.
To compare the safety of mexiletine PR vs mexiletine IR by assessing vital signs | Baseline to week 24
  To compare the safety of mexiletine PR vs mexiletine IR for the symptomatic treatment of myotonia in adult patients with non-dystrophic myotonias (myotonia congenita (MC), paramyotonia congenita (PC) and sodium channel myotonia (SCM)) by assessing vital signs. Vital signs will be obtained at each study visit and will include pulse, respiration, body temperature, and blood pressure. Unscheduled vital sign measurements may be obtained at the investigator's discretion during the study.
To compare the safety of mexiletine PR vs mexiletine IR by performing standard clinical laboratory evaluations | Baseline to week 24
  To compare the safety of mexiletine PR vs mexiletine IR for the symptomatic treatment of myotonia in adult patients with non-dystrophic myotonias (myotonia congenita (MC), paramyotonia congenita (PC) and sodium channel myotonia (SCM)) by performing standard clinical laboratory evaluations. Clinical laboratory samples will be collected under fasting conditions and hematology, serum chemistry, and urinalysis assessments will be performed

SECONDARY OUTCOMES:
Mean change in handgrip relaxation time | Baseline to week 24
  Opening Time (VHOT) functional evaluation by mean change in maximal voluntary isometric contraction (MVIC) and relaxation time by Video-recording of Hand. The dominant wrist and hand are placed on a bedside table with the forearm fully supinated. The patient is asked to open the hand after making a tight fist for 3-5 seconds 2 times within 30 minutes.
Mean change in health-related quality of life | Baseline to week 24
  Mean change in health-related quality of life (measured by INQoL) on a 7-point Likert scale
Mean change in MBS scores | Baseline to week 24
  Mean change in Myotonia Behavior Scale (MBS) scores on a 0-5 rating scale
Mean change in time to perform Timed-up and go (TUG) test | Baseline to week 24
  Mean change in time (seconds) to perform Timed-up and go (TUG) test
Mean change in VAS | Baseline to week 24
  Score for muscle stiffness (myotonia severity) as self-reported by patients on a Visual Analog Scale (VAS) on a 1-100 rating scale.
Mean change in Clinical Global Impression (CGI) - Efficacy Scale | Baseline to week 24
  Score for Clinical Global Impression (CGI) - Efficacy by a 5 rating scale of No Symptoms to Very Severe
Mean change in Clinical Global Impression (CGI) - Tolerability Index Scale | Baseline to week 24
  Mean change in Clinical Global Impression (CGI) - Tolerability Index Scale by a 7 rating scale of much worse to much better
Mean change in time to perform the 10-meter Walk Test | Baseline to week 24
  Mean change in time (seconds) to perform the 10-meter Walk Test (10mWT) 10mWT is a performance-based test assessing walking in two different conditions, own preferred speed and maximum speed, over a short distance. The time taken to walk 10 meters at usual comfortable and maximum speed is recorded with a stopwatch.
Mean change in Gastrointestinal function: The Gastroesophageal Reflux Disease-Health Related Quality of Life (GERD-HRQoL) | Baseline to week 24
  Mean change in Gastrointestinal function: The Gastroesophageal Reflux Disease-Health Related Quality of Life (GERD-HRQoL) by a 5 scale of no symptoms to Symptoms are incapacitating, unable to do daily activities
Mean change in CMRS Scale | Baseline to week 24
  Mean change in Clinical myotonia rating scale (CMRS)
Mean change Swallowing function | Baseline to week 24
  Mean change in Swallowing function: timed testing of swallowing
Preference between the two study treatments | Baseline to week 24
  Patients were also asked to give their preference between the 2 periods of treatment and to provide the primary reasons for their choice.

CONTACTS AND LOCATIONS:
Locations (1):
- Universitair Ziekenhuis Leuven"UZ Leuven Gasthuisberg Campus Herestraat 49 Leuven, 3000", Leuven, Belgium